CLINICAL TRIAL: NCT00829569
Title: Effects of Marine n-3 Fatty Acid Infusion on Insulin Sensitivity and Insulin Secretion in Type 2 Diabetes
Brief Title: n-3 Fatty Acid Infusion and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Norwegian Foundation for Health and Rehabilitation (Other); Novo Nordisk A/S (Industry); Norwegian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 4.2003.169; 03-14463 (Other: SLV); 15759 (Other: The Data Inspectorate); 03/05008 (Other: Biobank)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes
Keywords: Intralipid; Omegaven; fish oil; hyperinsulinemic isoglycemic clamps; C-peptide glucagon test; indirect calorimetry; F2-isoprostanes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intralipid with/without Omegaven (Experimental): Lipid infusion with/without marine n-3 fatty acids
  Interventions: Dietary Supplement: Intralipid +/- Omegaven

INTERVENTIONS:
Dietary Supplement: Intralipid +/- Omegaven — Intralipid®: the 500 ml 20% Intralipid will be infused during a hyperinsulinemic clamp. Infusion rate will increase from 50 to 100 ml/hour the first 30 min and then continue at 100 ml/hour for the next 210 min, infusion duration 240 min (4 hours) in all.
  Intralipid® + Omegaven®: In the 500 ml 20% Intralipid 100 ml will be replaced by 100 ml 10% Omegaven and infused during the hyperinsulinemic clamp as described for Intralipid only. Heparin (0.4 U/kg/min) will be added to both lipid emulsions.
  Content of marine n-3 fatty acids in 100 ml Omegaven will be 1.25-2.82 g EPA and 1.44-3.09 g DHA (seasoning variations of n-3 fatty acids in fish oil).
  Other Names: Fresenius Kabi, ATC main group B05B A 02; Intralipid Vnr 42 79 55; Omegaven Vnr 55 25 54

SUMMARY:
The purpose of this experimental study is to investigate whether an acute lipid infusion added marine n-3 fatty acids produces effects on insulin sensitivity in subjects with type 2 diabetes, when compared with an acute lipid infusion without marine n-3 fatty acids. Furthermore other effects on intermediary metabolism are tested for.

DETAILED DESCRIPTION:
Evidence indicates that n-3 fatty acids exert several beneficial effects. However, the effects of marine n-3 fatty acids on intermediary metabolism have not been completely elucidated. In a previous study of a high intake of marine n-3 fatty acids during 9 wk we demonstrated reduced insulin sensitivity and altered proportion of carbohydrate vs. fat oxidation in subjects with type 2 diabetes. These results question the use of high doses of n-3 supplements in type 2 diabetes. It is not known to what extent such effects in type 2 diabetes can be reproduced by intravenous administration of n-3 fatty acids and/or whether short term intravenous administration has other effects.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes defined by clinical criteria and by absence of antibodies to glutamic acid decarboxylase.
* HbA1c 5,5 - 8,5 %
* Blood pressure ≤ 170 mm Hg systolic and/or ≤ 105 mm Hg diastolic

Exclusion Criteria:

* insulin treatment
* hypertriglyceridemia (> 2,1 mmol/l TG)
* proliferative retinopathy, renal insufficiency (Se-Creatinine > 150 μmol/l)
* alcoholism, congestive heart failure or other serious diseases affecting the possibility of the subject to participate
* supplement with fish oil or marine n-3 fatty acids during the last 6 months before baseline
* Dicumarol treatment
* allergy to soya, fish or egg
* pregnancy or lactation
* smoking

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-01; Primary Completion 2004-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 4 hours

SECONDARY OUTCOMES:
n-3 fatty acid distribution | 4 hours
insulin secretion | 4 hours
energy metabolism | 4 hours
oxidative stress | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Valdemar Grill, M.D., Principal Investigator — St. Olavs Hospital, NTNU
Locations (1):
- Department of Medicine, Division of Endocrinology, St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Mostad IL, Bjerve KS, Basu S, Sutton P, Frayn KN, Grill V. Addition of n-3 fatty acids to a 4-hour lipid infusion does not affect insulin sensitivity, insulin secretion, or markers of oxidative stress in subjects with type 2 diabetes mellitus. Metabolism. 2009 Dec;58(12):1753-61. doi: 10.1016/j.metabol.2009.06.003. Epub 2009 Aug 27. PMID 19716144